CLINICAL TRIAL: NCT06902805
Title: Medium-and Long-term Efficacy of Two Ultrasound-guided Intra-articular Injections of onabotulinumtoxinA (Botox®) Combined With Custom-made Rigid Splinting in Painful Base-of-thumb Osteoarthritis : a Randomized Double-blind Controlled Trial in Three-parallel Arms
Brief Title: Efficacy of Two Ultrasound-guided Intra-articular Injections of Botox® Combined With Custom-made Rigid Splinting in Painful Base-of-thumb Osteoarthritis.
Acronym: RHIBOTII
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP230823
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Base-of-thumb Osteoarthritis; Osteoarthritis
Keywords: base-of-thumb osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 2 intra-articular injections of onabotulinumtoxinA (Experimental)
  Interventions: Drug: OnabotulinumtoxinA
- 1 intra-articular injection of onabotulinumtoxinA and 1 of normal saline (Experimental)
  Interventions: Drug: OnabotulinumtoxinA; Drug: Normal saline (placebo)
- 2 intra-articular injections of normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline (placebo)

INTERVENTIONS:
Drug: OnabotulinumtoxinA — intra-articular injection
  Arms: 1 intra-articular injection of onabotulinumtoxinA and 1 of normal saline; 2 intra-articular injections of onabotulinumtoxinA
Drug: Normal saline (placebo) — intra-articular injection
  Arms: 1 intra-articular injection of onabotulinumtoxinA and 1 of normal saline; 2 intra-articular injections of normal saline

SUMMARY:
The main objective of this study will be to compare the effects of 2 intra-articular injections of onabotulinumtoxinA with those of 1 intra-articular injection of onabotulinumtoxinA and 1 of normal saline and those of 2 intra-articular injections of normal saline on base-of-thumb pain at 6 months after the first injection.

DETAILED DESCRIPTION:
The base of the thumb is a frequent location of osteoarthritis. Base-of-thumb osteoarthritis affects middle-aged and older individuals and results in base-of-thumb pain and limitations in hand-specific activities. For the medium and long term, evidence suggests that splinting could reduce pain and improve hand function. For the short term, a combination of conservative treatments is recommended, with small-to-moderate treatment effect. However, use of intra-articular treatments (e.g., glucocorticoids and hyaluronan) for the short and medium term is currently debated. Use of intra-articular botulinum toxin A injection as a pain modulator in joint diseases has recently raised interest. Botulinum toxin A is a neurotoxin produced by Clostridium botulinum that inhibits acetylcholine release into the synaptic cleft in cholinergic nerve terminals. Additionally, treatment with botulinum toxin A showed intrinsic antinociceptive effects in various animal models of joint diseases.

In a pilot single-centred randomized controlled trial of 60 participants with painful base-of-thumb osteoarthritis, the investigators compared the effects of a single intra-articular injection of onabotulinumtoxinA (Botox® ) with those of a single intra-articular injection of normal saline on base-of-thumb pain, and found a significant reduction in pain.

Several perspectives raised from this pilot study. Like in the treatment of spasticity, repeated courses of intra-articular injections onabotulinumtoxinA may be necessary to obtain sustained analgesic effects over time. A replication of these findings in a multicentred setting, analysis of cost-effectiveness and description of safety at longer term are also needed before the official recommendation of this treatment. In RHIBOT II, the investigators hypothesize that 2 ultrasound-guided intra-articular injections of onabotulinumtoxinA, as an add-on therapy to custom-made rigid splinting, could reduce base-of-thumb pain at 6 months after the first injection.

ELIGIBILITY:
Inclusion Criteria:

* • Individuals aged at least 18 years;

  * Pain intensity of at least 30 on a self-administered 11-point pain numeric rating scale (0: no pain to 100: maximal pain);
  * Pain involving the base of the thumb;
  * X-ray evidence of trapezometacarpial osteoarthritis with at least two of the following items involving the trapezometacarpial joint: osteophytes, joint space narrowing, subchondral bone sclerosis, or subchondral cysts;
  * 1990 ACR classification criteria for hand osteoarthritis adapted to trapezometacarpial osteoarthritis.
  * Patient able to give written informed consent prior to participation in the study
  * Affiliation with a mode of social security (profit or being entitled).
  * Negative pregnancy test in women of childbearing potential

Exclusion Criteria:

* • Secondary osteoarthritis;

  * History of thumb surgery, inflammatory or crystal-associated rheumatic disease, or epilepsy;
  * Uncontrolled dysphagia, pneumonia, cardiovascular diseases, or clinical or subclinical signs of neuromuscular transmission disorders;
  * Contra-indication to onabotulinumtoxinA;
  * Neurological disorders involving the hands other than carpal tunnel syndrome;
  * Collagen disorders involving the hands;
  * Osteoarthritis predominating at the scaphotrapezial joint on x-ray;
  * Bilateral trapezometacarpial osteoarthritis without a predominant painful side;
  * Hand or wrist trauma for up to 2 months;
  * Intra-articular treatments for up to 2 months;
  * Use of IM, IV or oral corticosteroids for up to 2 months.
  * Protected adults (including individual under guardianship by court order)
  * Pregnant women and lactation; lack of contraception for women of childbearing potential
  * Patient participating in another investigational therapeutic study
  * Patient unable to speak and read french

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Base-of-thumb pain on a self-administered 11-point numeric rating scale | 6 months
  French version of the self-administered base-of-thumb pain numeric rating scale (0: no pain to 100: maximal pain)

SECONDARY OUTCOMES:
Base-of-thumb pain on a self-administered 11-point numeric rating scale | 1 and 12 months
  French version of the self-administered base-of-thumb pain numeric rating scale (0: no pain to 100: maximal pain)
Hand-specific activity limitations on the self-administered Cochin Hand Function Scale | 6 and 12 months
  mean change from baseline in hand-specific activity limitations in the previous 2 weeks on the self-administered Cochin Hand Function Scale (0: no limitations to 90: maximal limitations) at 6 and 12 months
patient global assessment on a self-administered 11-point numeric rating scale | 6 and 12 months
  mean change from baseline in patient global assessment on a self-administered 11-point numeric rating scale (0: worst possible condition to 100: best possible condition) at 6 and 12 months
health-related quality of life on the self-administered EQ-5D-5L questionnaire | 6 and 12 months
  mean change from baseline in health-related quality of life on the self-administered EQ-5D-5L questionnaire (0: death, 1: best quality of life) at 6 and 12 months
Osteoarthritis Research Society International-Outcome Measures in Rheumatology response | 6 and 12 months
  Osteoarthritis Research Society International-Outcome Measures in Rheumatology response (Response / No response)
estimated total costs and incremental cost-utility ratio | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christelle NGUYEN, MD,PhD, Principal Investigator — Organizational Affiliation: Université Paris Cité, Faculté de Santé | UFR de Médecine
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis du Pr François Rannou, Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No